CLINICAL TRIAL: NCT05604885
Title: A Two-part, Randomized, Double-blind, Multi-center, Placebo-controlled Study of the Dose-range, Safety and Efficacy of 4 and 12 Weeks of Treatment With AP1189 in Adult Rheumatoid Arthritis (RA) Patients With an Inadequate Response to Methotrexate (MTX) Alone - (RESOLVE)
Brief Title: A Dose-range Study of the Safety and Efficacy of Treatment in Adult Rheumatoid Arthritis Patients With an Inadequate Response to Methotrexate
Acronym: RESOLVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SynAct Pharma Aps (Industry)
Collaborators: NBCD A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SynAct-CS006
Record Dates: First submitted 2022-10-31; First posted 2022-11-03 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — N-(3-(1-(2-nitrophenyl)-1H-pyrrol-2-yl)allylidenamino)guanidine

STUDY DESIGN:
Intervention Model Description: Multi-center, two-part, randomized, double-blind, placebo-controlled study 4 and 12 weeks study with repeated doses of AP1189
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AP1189, 60 mg (Experimental): Part A: (AP1189, 60 mg); Part B: (TBD)
  Interventions: Drug: AP1189, 60 mg
- AP1189, 80 mg (Experimental): Part A: (AP1189, 80 mg); Part B: (TBD)
  Interventions: Drug: AP1189, 80 mg
- AP1189, 100 mg (Experimental): Part A: (AP1189, 100 mg); Part B: (TBD)
  Interventions: Drug: AP1189, 100 mg
- Placebo (Placebo Comparator): Part A: (placebo); Part B: (placebo).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AP1189, 60 mg — AP1189 tablets for oral use
  Arms: AP1189, 60 mg
Drug: AP1189, 80 mg — AP1189 tablets for oral use
  Arms: AP1189, 80 mg
Drug: AP1189, 100 mg — AP1189 tablets for oral use
  Arms: AP1189, 100 mg
Drug: Placebo — Matching placebo tablets for oral use
  Arms: Placebo

SUMMARY:
The RESOLVE study is a two-part, randomized, double-blind, multi-center, placebo-controlled study of the safety, dose-range finding confirmation, and efficacy of 4 (Part A) and 12 weeks (Part B) of treatment with AP1189 in adult RA patients with an inadequate response to MTX alone.

DETAILED DESCRIPTION:
In Part A approximately 120 randomized patients will be treated with either 60 mg AP1189, 80 mg AP1189, 100 mg AP1189 or placebo once daily for 4 weeks as add-on treatment to stable MTX treatment. Part A will conclude with an unblinded assessment for risk/benefit and a recommendation for dose selection for Part B.

In Part B patients will be randomized into groups of equal size evaluating 2-3 doses of AP1189 versus placebo. All doses will be administered once daily for 12 weeks as add-on treatment to stable MTX treatment. The proposed sample size per dose group/placebo group is 75 patients, by which the total study population of Part B may be either 225 or 300 patients, depending on the number of dose groups of AP1189 selected for evaluation based on Part A.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of RA according to the 2010 ACR/EULAR RA classification criteria and are ACR class I-III
* ≥6 swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts)
* Must meet at least one of the following parameters at Screening:

  1. A positive result for Anti-Cyclic Citrullinated Peptide (anti-CCP) or Rheumatoid Factor (RF),
  2. Serum CRP ≥ 6 mg/L based on central laboratory value
* Ongoing methotrexate therapy ≥12 weeks in a stable dose of 7.5 to 25 mg/week for at least 4 weeks prior to the baseline visit
* Subject has an inadequate clinical response to maximally tolerated methotrexate therapy
* Subjects should be receiving an adequate and prescribed stable dose of folic acid (≥5 mg/week total dose or as per local clinical practice) which should be confirmed or initiated at screening and continued throughout the study
* Negative QuantiFERON-in-Tube test (QFG-IT)
* Females of child-bearing potential must use of highly effective birth control method
* Male participant's partner must use highly effective birth control

Exclusion Criteria:

* Use of all other biologic or nonbiologic DMARDs and immunosuppressive therapy within 4 weeks prior to administration of the first dose of study drug
* Oral steroids at a dose >10 mg/day of prednisone or a prescription for oral steroids which has changed within 4 weeks of baseline
* Receipt of an intra-articular or parenteral corticosteroid injection within 4 weeks prior to baseline
* Major surgery (including joint operation) within 8 weeks prior to screening or planned surgery within the period of the study participation
* Rheumatic autoimmune disease other than RA
* Functional class IV as defined by the ACR Criteria for Classification of Functional Status in RA or wheelchair/bedbound
* Prior history of or current inflammatory joint disease other than RA
* Subjects with fibromyalgia
* Initiation or change in dose for NSAIDs (including low-dose aspirin and Cyclooxygenase (COX-2) inhibitors) within 2 weeks prior to baseline
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disease
* Serum Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) higher than 1.5 x the upper limit of normal (ULN) and alkaline phosphatase (ALP) and/or bilirubin values above the ULN at the screening visit
* Have prior renal transplant, current renal dialysis, or moderate to severe renal insufficiency
* Uncontrolled disease states, such as asthma, psoriasis, or inflammatory bowel disease where flares are commonly treated with oral or parenteral corticosteroids
* Evidence of active malignant disease (except basal cell carcinoma of the skin that has been excised and cured)
* History of alcohol, drug, or chemical abuse within the 6 months prior to screening
* Neuropathy or other painful, chronic conditions that might interfere with pain evaluation
* Body weight of >150 kg
* HBsAg positive and/or Anti-HBc with sign of current infection.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Part A: Change in ACR20 | 4 weeks
  The change in American College of Rheumatology 20% (ACR20) compared to baseline
Part B: Change in ACR20 | 12 weeks
  The change in American College of Rheumatology 20% (ACR20) compared to baseline
Number of reported Adverse Events | 12 weeks
  Evaluation of the safety and tolerability of AP1189 on the number and severity of reported Adverse Events, compared with placebo

SECONDARY OUTCOMES:
Part A: Change in ACR50 | 4 weeks
  The change in American College of Rheumatology 50% (ACR50) compared to baseline
Part B: Change in ACR50 | 12 weeks
  The change in American College of Rheumatology 50% (ACR50) compared to baseline
Part A: Change in ACR70 | 4 weeks
  The change in American College of Rheumatology 70% (ACR70) compared to baseline
Part B: Change in ACR70 | 12 weeks
  The change in American College of Rheumatology 70% (ACR70) compared to baseline
Part A: Change in CDAI | 4 weeks
  The change Clinical Disease Activity Index (CDAI) compared to baseline
Part B: Change in CDAI | 12 weeks
  The change Clinical Disease Activity Index (CDAI) compared to baseline
Part A: Change in DAS-28 | 4 weeks
  The change in Disease Activity Score (DAS-28), based on a C-Reactive Protein (CRP) value, compare to baseline
Part B: Change in DAS-28 | 12 weeks
  The change in Disease Activity Score (DAS-28), based on a C-Reactive Protein (CRP) value, compare to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Timofei Mosneaga Republican Clinical Hospital, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No